CLINICAL TRIAL: NCT02979730
Title: Proposal to Evaluate the Impact of Point of Care Liat Influenza A/B Testing in the Emergency Department at Boston Medical Center
Brief Title: Impact of Rapid Flu Testing in BMC ED
Acronym: FluProcess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Elissa Schechter-Perkins, Principal Investigator, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-35841
Record Dates: First submitted 2016-11-22; First posted 2016-12-02 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Influenza-Like Illness; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Lab Testing Arm (Active Comparator): For patients with clinical concern for influenza, the usual workflow in the BMC ED is that physicians order the collection of a nasopharyngeal swab (NPS) for influenza A/B testing to be performed in the core microbiology laboratory using one of two assays. The two influenza A/B-only assays available in the core lab are a) an instrumented fluorescent immunoassay rapid antigen test, the Sofia influenza A+B FIA (Quidel Corporation) and b) an automated real-time PCR test, the Xpert Flu (Cepheid, Inc.). Which test is ordered is at the discretion of the physician. Both the Sofia and Xpert assays provide a result callout to distinguish influenza type A from type B.
  Interventions: Other: Core Lab Test
- ED Point of Care Testing Arm (Experimental): Prior to the study the Cobas Liat Influenza A/B assay will be verified for patient care at BMC. The instrument and test kits will be available in the ED for use with study subjects randomized to this study arm. The Cobas Liat assay provides a result callout to distinguish influenza type A from type B.
  Interventions: Other: ED Point of Care Test

INTERVENTIONS:
Other: Core Lab Test — For patients randomized to the Core Lab Testing Arm, ED physicians will order an influenza test to be performed in the core lab.
  Arms: Core Lab Testing Arm
Other: ED Point of Care Test — For patients randomized to the ED Point of Care Testing Arm, the Research Assistant will perform influenza testing in the Emergency Department, using the Cobas Liat Influenza A/B assay
  Arms: ED Point of Care Testing Arm

SUMMARY:
The purpose of the study is to compare Emergency Department patients who undergo influenza testing using an FDA-approved point-of-care device (Cobas Liat Influenza A/B assay) located in the ED, to patients whose samples are sent to the BMC central laboratory. Patients who agree to participate will have their samples randomly assigned to be tested on either at the core lab, or on the POC device. The current turnaround time for samples sent to the laboratory is approximately two hours; investigators expect that the point of care device can reduce this time. Investigators will determine if the time to disposition and the administration of antibiotics is different in the group undergoing POC influenza testing compared to those undergoing laboratory-based influenza testing

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 21 years of age or older
* Presenting to the BMC main ED or Urgent Care area with influenza-like illness
* Physician ordered an influenza A/B diagnostic test

Exclusion Criteria:

* Previously enrolled in the study
* Any Influenza test result already available at the time approached by the ED RA
* Physician ordered comprehensive multiplex PCR respiratory pathogen assay instead of an initial influenza A/B-only test.
* Unable to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Time to Disposition | By the End of the ED visit (an average time of 4 hours)
  The time elapsed from when a patient was placed in the ED treatment room until the disposition (either admit, observe, or discharge) was ordered in the medical record

SECONDARY OUTCOMES:
Delivery of prescription or administration of antibiotics | by the end of ED visit (an average time of 4 hours)
  Whether patients either received a dose of antibiotics in the ED or received a prescription for antibiotics on discharge from the eD

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Perkins, MD, MPH, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No